CLINICAL TRIAL: NCT04437472
Title: Remote Collection of Patient Reported Toxicity Using SMS Text Messaging
Brief Title: Remote Collection of Patient Reported Toxicity Using SMS Text Messaging (CareSignal)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202005063
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CareSignal: -Participants will undergo a single training session on how to use the CareSignal software no more than 4 weeks before starting standard of care therapy. After the training session, patients will be encouraged by the treatment team to complete the baseline symptom report once they receive the questions via SMS prior to starting any therapy and to complete the weekly reports during therapy and in follow up.
  Interventions: Other: CareSignal

INTERVENTIONS:
Other: CareSignal — The CareSignal software will be programmed to automatically ask a subset of the NCI-PRO-CTCAE questions using SMS depending on patient group as designated by the treating physician: (1) thoracic radiation with chemotherapy, (2) thoracic radiation alone, (3) extremity/body wall sarcoma, and (4) other.

SUMMARY:
CareSignal has developed an application that allows for remote collection of patient-reported data such as symptoms or outcomes on any device compatible with the short message service (SMS), otherwise known as "text messaging". The software can be configured to complete symptom monitoring by surveying patients about toxicity using the PRO-CTCAE tools. PRO-CTCAE is the patient reported outcomes version of the CTCAE that was designed by the National Cancer Institute (NCI) for use in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Currently planning to receive radiotherapy for 2 or more fractions with or without chemotherapy.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Age 18 years or older.

Exclusion Criteria:

-Unable to reliably access and use a device compatible with CareSignal software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiation therapy at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Percentage of invited symptom reports completed during the study period | From treatment through 30 days follow-up (estimated to be 3 months)
Percentage of questions completed within each invited symptom report | From treatment through 30 days follow-up (estimated to be 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Spraker, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu